CLINICAL TRIAL: NCT01030601
Title: Analysis of the Effect of Intravitreal Dexamethasone Injection on Diabetic Macular Edema After Cataract Surgery (IDDMECS)
Acronym: IDDMECS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Michael Brent, MD, FRCSC, Toronto Western Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDDMECS
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Macular Edema; Pseudophakia
Keywords: Diabetic; Macular Edema; Pseudophakic; Dexamethasone; Intravitreal; Cataract surgery
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Pseudophakia | interventions — dexamethasone 21-phosphate

ARMS (2):
- Control (No Intervention): Diabetics undergoing routine cataract surgery
- Treatment (Experimental): Diabetics undergoing cataract surgery with injection of 0.5mg in 0.05cc of dexamethasone at the end of surgery
  Interventions: Drug: Dexamethasone sodium phosphate

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — 0.5mg in 0.05cc of Dexamethasone from a 10mg/ml vial
  Arms: Treatment

SUMMARY:
Macular Edema (Swelling of a particular site of the retina) can become a significant problem for Diabetics undergoing Cataract surgery. And a significant number of people who undergo Cataract surgery each year are diabetics. And when you multiply these two factors together you are left with a significant number of people who do not gain as much vision as their peers. Diabetics who develop Macular Edema actually can loose some vision after surgery and when you follow them up, they don't gain as much vision. This Study aims to prevent such an event from happening and therefore allow Diabetics to gain as much vision as they can from cataract surgery. This study will use Dexamethasone injected intravitreally (into the gel of the eye) at the end of cataract extraction to control Macular edema brought about by surgery. The main outcome is the central retina thickness and retinal volume as measured by Optical Coherence Tomography. Secondary outcomes are BCVA and incidence of Laser Treatment.

Other Drugs, life Bevacizumab and Pegaptanib, have been used for this purpose but they are expensive and have potential systemic side-effects due to anti-VEGF (vascular endothelial growth factor) actions. Dexamethasone has been used in the eye for decades and is short-lived, minimizing possible systemic effects. Moreover, this drug is at least 15x cheaper than the previously mentioned ones and therefore has tremendous benefit for developing countries. We seek an alternative drug that can reduce or prevent Macular edema at a less expensive and safer way.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients for Cataract Surgery with vision of ≤ 20/50 and > grade 3 any cataract type using the Lens Opacities Classification System III. Diabetics included must have at least one microaneurysm in the posterior pole (defined by the Superior and Inferior Arcade).

Exclusion Criteria:

* Without any diabetic retinopathy and those with active uncontrolled proliferative disease
* Retinal disease,other than Diabetes, that can affect macular edema
* Uveitis, a history of any other intraocular surgery or a history of uncontrolled glaucoma
* Eyes with cataract precluding proper OCT measurement pre-operatively
* Patients who will experience longer than usual operating time, complicated surgery, rupture of the posterior capsule, and iris or corneal burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Central Retinal Thickness | within 3 months after cataract surgery

SECONDARY OUTCOMES:
Best corrected visual acuity and incidence of laser treatments | within 3 months after cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Brent, MD, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada